CLINICAL TRIAL: NCT06677437
Title: Endovascular Preparation for Kidney Tranplantation
Acronym: EndoPreKiT
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_5431
Record Dates: First submitted 2024-06-17; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Renal Failure Chronic; Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single group of adult patients with chronic renal failure who are all awaiting a kidney transplant: This study focuses on a single group of adult patients with chronic renal failure who are all awaiting a kidney transplant, whether or not they are treated by extra-renal purification.
  These patients are contraindicated for transplantation due to their anatomical constraints: major arterial calcifications, iliac dissections, iliac stenoses and They can only receive the kidney transplant after arterial preparation.
  Interventions: Other: This is an observational and retrospective study

INTERVENTIONS:
Other: This is an observational and retrospective study — It concerns all patients with chronic renal failure awaiting a kidney transplant, and presenting a contraindication to the transplant due to their anatomical constraints: major arterial calcifications, iliac dissections, iliac stenoses. They can only receive the kidney transplant after arterial preparation. These patients will be included and will benefit from endovascular preparation for the kidney transplant using a tailor-made arterial stent.
  Imaging examinations and follow-up clinical data will be analyzed. Reinterventions and causes of death will be analyzed.
  An information sheet will be given to patients; if the patient refuses the use of their data, it will not be collected.
  Data collection will be carried out by ARCs or PIs of the centers from medical records. The data will be pseudo-anonymized, entered into a REDCAP database shared between each center.

SUMMARY:
This national study is a feasibility study. It wants to validate all stages of the endovascular preparation of the iliac axis up to the kidney transplant for patients in whom the installation of a tailor-made endoprosthesis was necessary beforehand.

These patients are currently at a therapeutic impasse. This strategy of renal transplantation on an iliac artery endoprosthesis could ultimately give them access to the transplant with an improvement in quality of life and survival, for lower costs of care for the hospital and safety. less social than treatment by hemodialysis

ELIGIBILITY:
Inclusion Criteria:

1. Patient from 18 to 85 years old (beyond 85 years old, guidance must remain exceptional)
2. Patients with chronic renal failure
3. Waiting for a kidney transplant
4. Who have a vascular contraindication to renal transplantation because of their anatomical constraints.

Exclusion Criteria:

1-All criteria contraindicating kidney transplant other than for arterial anatomical problems: All criteria contraindicating kidney transplant other than for arterial anatomical problems:

* A progressive cancer, which is not cured,
* An uncontrolled infectious disease,
* Severe cardiovascular or respiratory disease making general anesthesia impossible,
* Unstabilized psychiatric disorders or illness,
* Dementia proven to have progressed after specialist advice
* Major obesity, with a body mass index greater than 50 kg/m2
* Patient refusal 2. Patient under curatorship 3. Pregnant woman 4. Patients for whom it will not be possible to organize regular medical follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns adult patients with chronic renal failure who are all awaiting a kidney transplant, whether or not they are treated by extra-renal purification.
  These patients are contraindicated for transplantation due to their anatomical constraints: major arterial calcifications, iliac dissections, iliac stenoses and They can only receive the kidney transplant after arterial preparation.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the success of endovascular arterial preparation for grafting Renal. | "From enrollment to the end of treatment at 12 months
  The success of arterial preparation for renal transplantation will be evaluated by:
  * Collect safety estimators, absence of serious complications (hemorrhage, acute/subacute ischemia of the lower limb, death, serious post-operative cardiorespiratory event, failure of renal function for non-dialysis patients) Validity at 1 month of an endovascular preparation for renal transplantation by tailor-made arterial stent by the success of the installation, the absence of endoleak and the good anteroposterior positioning of the stent
  * Effectiveness at 1 month of endovascular preparation for renal transplantation by tailor-made arterial stent by permeability confirmed by Doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- HCL Hopital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No